CLINICAL TRIAL: NCT06434233
Title: A Randomized Control Trial for Opioid Use After Laparoscopic Salpingectomy
Brief Title: Opioid Use After Laparoscopic Salpingectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00308549
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use; Post-operative Pain; Sterility, Female
MeSH Terms: conditions — Pain, Postoperative; Infertility, Female | interventions — Acetaminophen; Ibuprofen; Oxycodone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Opioid Post-Op Pain Regimen (Active Comparator): Patients randomized to Arm 1 will receive the current most commonly prescribed pain control regimen after a minimally invasive tubal sterilization procedure at discharge.
  These medications include:
  Tylenol 500 mg orally every 6 hours scheduled x 30 tablets Ibuprofen 600 mg orally every 6 hours scheduled x 30 tablets and Oxycodone 5 mg orally every 4 hours as needed x 12 tablets
  All patients will be instructed to use Acetaminophen and Ibuprofen around the clock for the first 72 hours and as needed thereafter
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen; Drug: Oxycodone
- Arm 2 - Non-Opioid Post-Op Pain Regimen (Experimental): Patients randomized to Arm 2 will not receive an opioid prescription after minimally invasive tubal sterilization procedures at discharge. They will receive only Tylenol and Ibuprofen as follows:
  Tylenol 500 mg orally every 6 hours scheduled x 30 tablets Ibuprofen 600 mg orally every 6 hours scheduled x 30 tablets and
  All patients will be instructed to use Acetaminophen and Ibuprofen around the clock for the first 72 hours and as needed thereafter.
  Participants will be informed that if they need additional pain medications, these will not be withheld. Participants in the second arm who require additional pain medications will receive the same amount of oxycodone as in arm 1.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — All patients will receive Acetaminophen 500 mg orally every 6 hours scheduled x 30 tablets at post-operative discharge.
  All patients will be instructed to take Acetaminophen around the clock for the first 72 hours and as needed thereafter.
  Other Names: Tylenol
Drug: Ibuprofen — All patients will receive Ibuprofen 600 mg orally every 6 hours scheduled x 30 tablets at post-operative discharge.
  All patients will be instructed to take Ibuprofen around the clock for the first 72 hours and as needed thereafter.
Drug: Oxycodone — Patients randomized to Arm 1 will receive Oxycodone 5 mg orally every 4 hours as needed x 12 tablets at post-operative discharge
  Patients randomized to Arm 2 will not receive an Oxycodone prescription at post-operative discharge.
  However, participants will be informed that if they need additional pain medications, these will not be withheld. Participants in the second arm who require additional pain medications will receive the same amount of Oxycodone as in arm 1
  Arms: Arm 1 - Opioid Post-Op Pain Regimen

SUMMARY:
The purpose of this study is to evaluate patient-reported post-operative pain scores following minimally invasive tubal sterilization procedures to determine if a multimodal, non-opioid pain control regimen is non-inferior to a pain control regimen including opioids.

The study team hypothesizes that with extensive counseling on pain management, multimodal medication use, and expectation with non-opioid methods can effectively eliminate the need for opioid prescriptions after laparoscopic salpingectomy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a fallopian tube (unilateral and/or bilateral)
* Age 18 years old and above
* Undergoing minimally invasive (laparoscopic or robotic) unilateral or bilateral salpingectomy or other tubal sterilization procedure as the primary procedure
* Benign indications for salpingectomy/tubal sterilization
* Agreeing to participate

Exclusion Criteria:

* Chronic pain syndromes patients including fibromyalgia
* Patients currently on long-term (i.e. for more than three months) opioid use
* Conversion to laparotomy
* Allergy or other contraindication to the prescribed medications such as acetaminophen or oxycodone
* Salpingectomy that occurs in conjunction with a major Gyn surgery (i.e. hysterectomy, etc)
* Salpingectomy performed for treatment of ectopic pregnancy
* Patients with a history of gastritis and/or GI bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Numeric post-operative pain score | post-operative day 1 and post-operative day 7
  Patient reported pain on "Post-Operative Day 1 Survey" and "Post-Operative Day 7 Survey" using the Likert pain scale from 0 to 10, where 0 is no pain and 10 is severe pain. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Satisfaction with post-operative pain relief | post-operative day 1 and post-operative day 7
  As indicated on "Post-Operative Day 1 Survey" and "Post-Operative Day 7 Survey" by a binary "yes" or "no" response. "Yes" indicates a favorable outcome and "no" indicates a worse outcome.
Satisfaction with post-operative mobility | post-operative day 1 and post-operative day 7
  As indicated on "Post-Operative Day 1 Survey" and "Post-Operative Day 7 Survey" by a binary "yes" or "no" response. "Yes" indicates a favorable outcome and "no" indicates a worse outcome.
Total narcotic consumption at one week post-operative | post-operative day 7
  Number of Oxycodone pills used by each patient by the end of post-operative day 7
Occurrence of defined opioid related side effects (N/V, constipation, dizziness, itchiness) | post-operative day 1 and post-operative day 7
  As indicated on "Post-Operative Day 1 Survey" and "Post-Operative Day 7 Survey" by a binary "yes" or "no" response. "No" indicates a favorable outcome and "yes" indicates a worse outcome.
Suboptimal pain control as assessed by the number of patients requesting additional medication or seeking unplanned medical care for a post-surgical pain-related concern | Within 30 days of surgery
  Number of patients who request additional pain medications at the time of post-operative surveys, call provider phone line for additional pain medications, or return to an Emergency Department, clinic/office, etc due to a pain related issue.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Borahay, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States